CLINICAL TRIAL: NCT03297723
Title: Effectiveness of a Patient Therapeutic Education Program in Improving Pain Management
Acronym: EFFADOL-K
Status: Completed | Type: Observational
Sponsor: Centre Francois Baclesse (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2016-A01405-46
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2023-07

CONDITIONS: Pain Cancer
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental arm: The experimental group will be constituted after the medical staff was trained to TPE. Cancer patients will benefit from a PEP aiming at learning how to better manage their pain.
  Interventions: Other: Therapeutic education Programm
- Controle arm: The control group will be constituted before the training of the medical staff to TPE. Patients' pain will be managed conventionally.

INTERVENTIONS:
Other: Therapeutic education Programm — Intervention will include:
  * an identification of educational needs and expectations,
  * a bilateral agreement between patient and medical staff on the priority skills acquirement,
  * a structured educational activities tailored to the patient's need.
  * the making of an educational record.
  Groups: Experimental arm

SUMMARY:
Pain is one of the most feared and burdensome symptoms experienced by cancer patients. Its prevalence has been estimated by INCa1 in 2012 at 48% in patients undergoing cancer treatment, and unrelieved pain is directly associated with significantly reduced quality of life (QoL)2. A large part of cancer pain undertreatment can be attributed to patient-related barriers. Patient barriers are multifactorial and often result from a lack of knowledge about cancer pain and its self-management. They mainly consist of misconceptions about opioids and their side effects, nonadherence, and reluctance to alert health care providers to unrelieved pain. Patient education enables people with chronic disease to manage their illness, and has been considered in the field of cancer research as an important strategy to achieve optimal pain control.

In Basse-Normandie french region, the "Health Regional Plan, pain aspect" has identified the theme " pain education program " as a priority.

The main endpoint is the decrease of pain interference with daily life (using the Brief Pain Inventory). The experimental group, consisting of cancer pain patients, will benefit from the education program by previously trained health care providers. It will be compared with the control group, consisting with patients whose pain will be conventionally managed before the professional training in therapeutic education.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from a cancer which diagnosis has been established since at least 1 month
* Patient who suffers from pain related to the pathology or its treatment:
* receiving an analgesic treatment since at least 1 month
* moderate to severe pain intensity in the previous week : average pain score greater than 4 (on a 0-10 numerical rating scale), OR pain leading to insomnia OR 4 daily breakthrough pain, which interferes with daily activities
* Patient with a life expectancy > or = 6 months
* Health compatible with the PEP requirements (WHO performance scale > or = 2)
* Patient v 18 years old
* Patient able to understand, speak and read French
* Patient without cognitive dysfunctions
* Patient with a signed informed consent before inclusion in the study

Exclusion Criteria:

* Primary central nervous system or cerebral metastases
* Disorders of higher functions documented
* Evolutionary psychiatric pathology
* Drug user
* Abuse of alcohol exceeding WHO recommendations
* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient suffering from a cancer and suffering from pain
Sampling Method: Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
the decrease of pain impact on daily life activities based on a decrease of 2 points (on a 0-10 scale) between mean values measured before and after the PEP (at 1 month). | 1 month

SECONDARY OUTCOMES:
The proportion of patients adhering to the full ETP program (3 workshops), | 1 month

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - centre Hospitalier d'Alençon, Alençon
  - Centre Hospitalier d'Argentan, Argentan
  - Centre Hospitalier AVRANCHES-GRANVILLE, Avranches
  - Centre Hospitalier Bayeux, Bayeux
  - Centre François Baclesse, Caen
  - CHU CAEN, Caen
  - Hopital privé Paul d'Egine, Champigny-sur-Marne
  - Centre Hospitalier de Cherbourg, Cherbourg-Octeville
  - Ch Dieppe, Dieppe
  - Centre Hospitalier de Flers, Flers
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier Lisieux, Lisieux
  - Hopital Européen Georges Pompidou (HEGP), Paris
  - Centre Hospitalier de Saint-lo, Saint-Lô
  - Ghpso Senlis, Senlis
  - IGR, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prevost V, Delorme C, Leconte A, Le Chevalier A, Fourel L, Gicquere M, Grach MC, Le Caer F, Clarisse B. Cancer Pain and Patient Education: Strategy, Implementation, Difficulties and Opportunities of EFFADOL, a Regional Collaborative Programme. J Cancer Educ. 2022 Aug;37(4):1089-1098. doi: 10.1007/s13187-020-01924-w. Epub 2020 Nov 19. PMID 33215294
- [Derived] Prevost V, Heutte N, Leconte A, Licaj I, Delorme C, Clarisse B; EFFADOL-Group. Effectiveness of a therapeutic patient education program in improving cancer pain management: EFFADOL, a stepped-wedge randomised controlled trial. BMC Cancer. 2019 Jul 8;19(1):673. doi: 10.1186/s12885-019-5836-5. PMID 31286871